CLINICAL TRIAL: NCT07299890
Title: An Exploratory Study of Pertuzumab and Trastuzumab in Combination With Palbociclib and Exemestane as Neoadjuvant Therapy for Triple-Positive Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yue-Yin Pan, chief physicians, Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-LLYJ-0008
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; palbociclib; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Trastuzumab and Pertuzumab Combination with Palbociclib and Exemestane
  Interventions: Drug: Trastuzumab and Pertuzumab Combination with Palbociclib and Exemestane

INTERVENTIONS:
Drug: Trastuzumab and Pertuzumab Combination with Palbociclib and Exemestane — Neoadjuvant treatment regimen:
  QL1701 (Trastuzumab for Injection): First dose 8mg/kg, then 6mg/kg, every 3 weeks, for a total of 6 cycles; QL1209 (Pertuzumab Injection): First dose 840mg, then 420mg, every 3 weeks, for a total of 6 cycles; Palbociclib: 125mg/day, days 1-21, every 4 weeks, for a total of 5 cycles; Exemestane: 25mg/day, every 4 weeks, for a total of 5 cycles.

SUMMARY:
This study is a prospective, multicenter, single-arm, exploratory study. A total of 90 patients with early/later-stage triple-positive breast cancer who were scheduled to receive neoadjuvant therapy were recruited. They received neoadjuvant treatment with trastuzumab, pertuzumab, palbociclib, and exemestane in combination. The aim of this study is to evaluate the efficacy and safety of the neoadjuvant treatment regimen of trastuzumab-pertuzumab combined with palbociclib and exemestane in triple-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient must meet all of the following criteria to be included in the study:

  1. The tumor stage must be in accordance with the 8th edition of the AJCC standard, being stage II-III for the initial diagnosis;
  2. Pre-menopausal or perimenopausal patients (if this is the case, combined with OFS, which includes bilateral oophorectomy or GnRHa drugs), or post-menopausal patients;
  3. All patients must have been pathologically confirmed as HR+/HER2 receptor positive. The estrogen receptor (ER) is positive (>10%), the progesterone receptor (PR) is positive (>1%), and the HER2 receptor is positive. Follow the 2018 ASCO-CAP HER2 positive interpretation guideline standards. The immunohistochemistry (IHC) score is 3+ or 2+ and the in situ hybridization (ISH) test is positive (ISH amplification rate ≥ 2.0);
  4. Age 18-75 years (inclusive of 18 and 75), female;
  5. ECOG score 0-1;
  6. Expected survival time ≥ 12 weeks;
  7. According to the RECIST 1.1 standard, there must be at least one measurable lesion;
  8. The functional level of organs must meet the following requirements: (a) Blood routine: ANC ≥ 1.5×109/L; PLT ≥ 90×109/L; Hb ≥ 90g/L; (b) Blood biochemistry: TBIL ≤ 1.5×ULN; ALT and AST ≤ 3×ULN; BUN and Cr ≤ 1.5×ULN and creatinine clearance rate ≥ 50 mL/min; (c) Cardiac echocardiography: Left ventricular ejection fraction ≥ 50%:
  9. The subject voluntarily joins this study, signs the informed consent, has good compliance and is willing to cooperate with follow-up.

Exclusion Criteria:

* If the patient meets any of the following conditions, they will not be eligible:

  1. Has received any form of anti-tumor treatment (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.);
  2. Is concurrently receiving other anti-tumor drug treatments;
  3. Stage IV breast cancer;
  4. Breast cancer without pathological tissue diagnosis;
  5. Has had other malignant tumors within the past 5 years, except for cured cervical carcinoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin;
  6. Patients with severe dysfunction of important organs such as heart, liver, and kidney;
  7. Unable to swallow, chronic diarrhea and intestinal obstruction, with multiple factors affecting the administration and absorption of the drugs;
  8. Participated in other drug clinical trials within 4 weeks before enrollment;
  9. Has a history of immunodeficiency diseases, including positive HIV test, HCV, active viral hepatitis or other acquired or congenital immune deficiency diseases, or a history of organ transplantation;
  10. Has a known history of allergic reaction to the components of this drug regimen;
  11. Has had any heart diseases, including: requiring drug treatment or clinically significant arrhythmia; myocardial infarction; heart failure; any other heart diseases judged by the researcher as unsuitable for participation in this trial;
  12. Pregnant or lactating female patients, female patients with reproductive capacity and positive baseline pregnancy test results;
  13. According to the investigator's judgment, there are serious accompanying diseases that endanger the patient's safety or affect the patient's completion of the study (including but not limited to severe hypertension that cannot be controlled by drugs, severe diabetes, active infection, etc.);
  14. Has a clear history of neurological or mental disorders, including epilepsy or dementia;
  15. The investigator considers that the patient is not suitable for participating in this study in any other circumstances.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
tpCR rate，total physiological complex response | From the time of enrollment to one month after the surgery
  After the resection of the primary tumor, microscopic examination of the breast and the ipsilateral axillary lymph nodes revealed no invasive tumor cells (ypT0/is ypN0)

SECONDARY OUTCOMES:
bpCR，breast physiological complex response | From the time of enrollment to one month after the surgery
  After the primary tumor was removed, microscopic examination of the breast revealed no invasive tumor cells (ypT0/is)
The proportion of patients with Miller & Payne classification (MP classification) at grades 4 to 5 | From the time of enrollment to one month after the surgery
EFS，Event-free survival | baseline，1year，up to 2year
  The time from the start of medication to the occurrence of any of the following events for the first time: disease progression making surgical treatment impossible, local or distant recurrence, death due to any cause, etc.
ORR，Objective Response Rate | 6-12 months
  The proportion of patients whose tumor volume has decreased by 30% and has remained stable for more than four weeks is referred to as the sum of complete response (CR) and partial response (PR).
OS，Overall Survival | baseline，1year，up to 2year
  Refers to the period from the start of medication use until death occurs due to any cause.
adverse event | up to 2year
  Collect all adverse events that occurred in all subjects from the signing of the informed consent to 28 days after the cessation of medication, including clinical symptoms and abnormal vital signs, as well as abnormalities in laboratory tests. Record the clinical manifestations, severity, occurrence time, duration, treatment methods, prognosis, and determine the correlation between these events and the test drug.
PRO | through study completion, an average of 1 year
  Outcome indicators reported by the patients，Score using the Chinese version of the EORTC Quality of Life Questionnaire Core 30 (QLQ-C30, V3.0)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol